CLINICAL TRIAL: NCT01044680
Title: The Effects of NUTRIOSE®FB Dietary Fiber Supplementation on the Satiety, Body Fat Distribution, and Metabolic Syndrome Biomarkers of Overweight Adult Chinese Men 20-35 Years of Age.
Brief Title: Effects of NUTRIOSE®FB Dietary Fiber Supplementation on Satiety, Body Fat, and Metabolic Syndrome in Overweight Adult Men
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Roquette Freres (Industry)
Collaborators: Sprim Advanced Life Sciences (Other)
Responsible Party: Laetitia Guerin-Deremaux, Roquette Freres
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 06-10- CN-Roquette-01
Record Dates: First submitted 2010-01-06; First posted 2010-01-08 (Estimated); Last update posted 2010-01-08 (Estimated); Status verified 2010-01

CONDITIONS: Overweight; Metabolic Syndrome X
Keywords: fiber; metabolic syndrome; overweight; satiety
MeSH Terms: conditions — Overweight; Metabolic Syndrome | interventions — NUTRIOSE

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutriose (Experimental): 17 g NUTRIOSE consumed twice daily for 12 weeks
  Interventions: Dietary Supplement: NUTRIOSE
- Placebo (Placebo Comparator): 17 g maltodextrin consumed twice daily for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: NUTRIOSE — 17 grams of NUTRIOSE consumed twice daily for 12 weeks
  Arms: Nutriose
Dietary Supplement: Placebo — 17 g maltodextrin consumed twice daily for 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study was to determine the effects of NUTRIOSE® supplementation on body composition, satiety, and determinants of metabolic syndrome in overweight men.

DETAILED DESCRIPTION:
Previous trials of fiber supplementation have yielded equivocal results on body composition, satiety, and determinants of metabolic syndrome. This double-blind, randomized, placebo-controlled study was conducted to determine the effects of a proprietary soluble dextrin dietary fiber supplement (NUTRIOSE®) on these parameters in overweight males.

ELIGIBILITY:
Inclusion Criteria:

* males 20-35 years
* body mass index of 24-28 kg/m2
* current employment and residence at one of three manufacturing plants with a controlled setting and with similar regimented working conditions 7 days a week

Exclusion Criteria:

* current or recent dietary fiber supplementation
* use of lipid-lowering/hypertension medication
* current insulin injection use
* contraindication to fiber supplements, e.g. Crohn's disease
* allergy to wheat products
* recent or current antibiotic use

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2006-10; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Determinants of metabolic syndrome | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shuguang Li, MD, Principal Investigator — Tongji University Medical College
Locations (1):
- Tongji University Medical College, Shanghai, China

REFERENCES:
- [Background] Pasman W, Wils D, Saniez MH, Kardinaal A. Long-term gastrointestinal tolerance of NUTRIOSE FB in healthy men. Eur J Clin Nutr. 2006 Aug;60(8):1024-34. doi: 10.1038/sj.ejcn.1602418. Epub 2006 Feb 15. PMID 16482066
- [Background] van den Heuvel EG, Wils D, Pasman WJ, Saniez MH, Kardinaal AF. Dietary supplementation of different doses of NUTRIOSE FB, a fermentable dextrin, alters the activity of faecal enzymes in healthy men. Eur J Nutr. 2005 Oct;44(7):445-51. doi: 10.1007/s00394-005-0552-0. Epub 2005 Feb 9. PMID 15696402
- [Background] van den Heuvel EG, Wils D, Pasman WJ, Bakker M, Saniez MH, Kardinaal AF. Short-term digestive tolerance of different doses of NUTRIOSE FB, a food dextrin, in adult men. Eur J Clin Nutr. 2004 Jul;58(7):1046-55. doi: 10.1038/sj.ejcn.1601930. PMID 15220947
- [Derived] Li S, Guerin-Deremaux L, Pochat M, Wils D, Reifer C, Miller LE. NUTRIOSE dietary fiber supplementation improves insulin resistance and determinants of metabolic syndrome in overweight men: a double-blind, randomized, placebo-controlled study. Appl Physiol Nutr Metab. 2010 Dec;35(6):773-82. doi: 10.1139/H10-074. PMID 21164548